CLINICAL TRIAL: NCT03514446
Title: Efficacy of Seven and Fourteen Days of Antibiotic Treatment in Uncomplicated Staphylococcus Aureus Bacteremia: A Randomized, Non-blinded, Non-inferiority Interventional Study
Brief Title: Seven Versus Fourteen Days of Treatment in Uncomplicated Staphylococcus Aureus Bacteremia
Acronym: SAB7
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, Clinical Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-17027414; 2017-003529-13 (EudraCT Number)
Record Dates: First submitted 2017-11-10; First posted 2018-05-02 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Staphylococcus Aureus Bacteremia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antibiotic therapy duration for 7 days (Experimental)
  Interventions: Drug: Antibiotic therapy duration for 7 days
- Antibiotic therapy duration for 14 days (No Intervention)

INTERVENTIONS:
Drug: Antibiotic therapy duration for 7 days — Antibiotic therapy for seven days
  Arms: Antibiotic therapy duration for 7 days

SUMMARY:
Introduction: Staphylococcus aureus bacteremia (SAB) plays an important role in long-course antibiotic therapy. Current international guidelines recommend fourteen days of intravenous antibiotic treatment for SAB in order to minimize risks of secondary deep infections and complications. However, patients with simple SAB are known to have a low risk of complications. Reducing treatment length in uncomplicated SAB would reduce the total consumption of antibiotics, adverse events and duration of hospital admission. SAB7 seeks to determine if seven days of antibiotic treatment in patients with uncomplicated SAB is non-inferior to fourteen days of treatment.

Method: The study is designed as a randomized, non-blinded, non-inferiority interventional study. Primary measure of outcome will be failure to treatment or recurrence of SAB twelve weeks after termination of antibiotic treatment. As a measure of secondary outcome the prevalence of severe adverse effects will be evaluated, in particular secondary infection with Clostridium difficile, mortality as well as public health related costs. Patients identified with uncomplicated SAB, are randomized 1:1 in two parallel arms to seven or fourteen days of antimicrobial treatment, respectively. Endpoints will be tested with a statistical non-inferiority margin of 10%.

Conclusion: SAB 7 will determine if seven days of antibiotic treatment in patients with uncomplicated SAB is sufficient and safe, potentially modifying current treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Blood culture positive for Staphylococcus aureus
* Antibiotic treatment with antimicrobial activity to S. aureus administrated within 12 hours of the first positive blood culture
* Temperature < 37,5 degrees celsius at randomization
* S. aureus negative follow-up blood culture obtained 48-96 hours after microbiological verified SAB.
* Patients written consent obtained

Exclusion Criteria:

* Persistence of S. aureus bacteremia before randomization (S. aureus positive follow-up blood culture obtained 48-96 hours of the first positive blood culture)
* Polymicrobial infection
* Antibiotic treatment whit no antimicrobial activity to S. aureus administrated more than 12 hours of the first positive blood culture
* Endocarditis or other intracardiac infection demonstrated with transthoracic or transesophageal echocardiography
* Previous history of endocarditis
* Pacemaker or other intracardiac implant
* Failure to remove a likely focus of infection, such as central venous catheter within 72 hours of the first positive blood culture.
* Prosthetics in joints and bones or vascular grafts
* Pneumonia or infection involving bone or joints
* Previously bone/join infection
* S. aureus infection within the last 90 days
* Pregnancy or breastfeeding
* Neutropenia (blood neutrophils < 1,0 x 109/l)
* Untreated cancer
* Chemotherapy within 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
90-day survival without clinical or microbiological failure to treatment or relapse | up to 90 days

SECONDARY OUTCOMES:
Microbiologically failure to treatment | less than 7 days after treatment termination
  Verified S. aureus infection of the same genotype as the initial infection
Microbiologically relapse | more than 7 days after treatment termination
  Verified S. aureus infection of the same genotype as the initial infection
Clinical failure to treatment or relapse | Up to day 90
  Initiation of anti-staphylococcal therapy for more than 48 hours due to suspected recurrence.
Mortality | Days 14, 28, 90 and 180
  All-cause mortality
Severe adverse events | Up to 26 weeks
  grade 3 or above adverse events
Acute renal injury | Up to 26 weeks
  A 1.5 fold increase in creatinine or a 25% decrease of the glomerular filtration rate (GFR)
Clostridium difficile infection | Up to 26 weeks
  Microbiologically verified C. difficile infection
Multidrug-resistance organism | Up to 26 weeks
  Microbiologically verified multidrug-resistance organism
Health-associated costs | Up to 26 weeks
  Public health related cost estimated from a general consideration of the expenses associated with hospitalization for SAB.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banaei N, Anikst V, Schroeder LF. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Jun 11;372(24):2368-9. doi: 10.1056/NEJMc1505190. No abstract available. PMID 26061852
- [Background] Kaasch AJ, Fatkenheuer G, Prinz-Langenohl R, Paulus U, Hellmich M, Weiss V, Jung N, Rieg S, Kern WV, Seifert H; SABATO trial group (with linked authorship to the individuals in the Acknowledgements section). Early oral switch therapy in low-risk Staphylococcus aureus bloodstream infection (SABATO): study protocol for a randomized controlled trial. Trials. 2015 Oct 9;16:450. doi: 10.1186/s13063-015-0973-x. PMID 26452342
- [Background] Thwaites GE, Edgeworth JD, Gkrania-Klotsas E, Kirby A, Tilley R, Torok ME, Walker S, Wertheim HF, Wilson P, Llewelyn MJ; UK Clinical Infection Research Group. Clinical management of Staphylococcus aureus bacteraemia. Lancet Infect Dis. 2011 Mar;11(3):208-22. doi: 10.1016/S1473-3099(10)70285-1. PMID 21371655
- [Background] Blyth CC, Darragh H, Whelan A, O'Shea JP, Beaman MH, McCarthy JS. Evaluation of clinical guidelines for the management of Staphylococcus aureus bacteraemia. Intern Med J. 2002 May-Jun;32(5-6):224-32. doi: 10.1046/j.1445-5994.2001.00205.x. PMID 12036220
- [Background] Benfield T, Espersen F, Frimodt-Moller N, Jensen AG, Larsen AR, Pallesen LV, Skov R, Westh H, Skinhoj P. Increasing incidence but decreasing in-hospital mortality of adult Staphylococcus aureus bacteraemia between 1981 and 2000. Clin Microbiol Infect. 2007 Mar;13(3):257-63. doi: 10.1111/j.1469-0691.2006.01589.x. PMID 17391379
- [Background] Zeylemaker MM, Jaspers CA, van Kraaij MG, Visser MR, Hoepelman IM. Long-term infectious complications and their relation to treatment duration in catheter-related Staphylococcus aureus bacteremia. Eur J Clin Microbiol Infect Dis. 2001 Jun;20(6):380-4. doi: 10.1007/pl00011278. PMID 11476436
- [Background] Raad II, Sabbagh MF. Optimal duration of therapy for catheter-related Staphylococcus aureus bacteremia: a study of 55 cases and review. Clin Infect Dis. 1992 Jan;14(1):75-82. doi: 10.1093/clinids/14.1.75. PMID 1571466
- [Background] Fowler VG Jr, Sanders LL, Sexton DJ, Kong L, Marr KA, Gopal AK, Gottlieb G, McClelland RS, Corey GR. Outcome of Staphylococcus aureus bacteremia according to compliance with recommendations of infectious diseases specialists: experience with 244 patients. Clin Infect Dis. 1998 Sep;27(3):478-86. doi: 10.1086/514686. PMID 9770144
- [Background] Mylotte JM, McDermott C, Spooner JA. Prospective study of 114 consecutive episodes of Staphylococcus aureus bacteremia. Rev Infect Dis. 1987 Sep-Oct;9(5):891-907. doi: 10.1093/clinids/9.5.891. PMID 3317734
- [Background] Ehni WF, Reller LB. Short-course therapy for catheter-associated Staphylococcus aureus bacteremia. Arch Intern Med. 1989 Mar;149(3):533-6. PMID 2919931
- [Background] Larsen AR, Stegger M, Sorum M. spa typing directly from a mecA, spa and pvl multiplex PCR assay-a cost-effective improvement for methicillin-resistant Staphylococcus aureus surveillance. Clin Microbiol Infect. 2008 Jun;14(6):611-4. doi: 10.1111/j.1469-0691.2008.01995.x. Epub 2008 Apr 3. PMID 18393997
- [Background] Mejer N, Westh H, Schonheyder HC, Jensen AG, Larsen AR, Skov R, Benfield T; Danish Staphylococcal Bacteraemia Study Group. Stable incidence and continued improvement in short term mortality of Staphylococcus aureus bacteraemia between 1995 and 2008. BMC Infect Dis. 2012 Oct 17;12:260. doi: 10.1186/1471-2334-12-260. PMID 23075215
- [Background] Mylotte JM, McDermott C. Staphylococcus aureus bacteremia caused by infected intravenous catheters. Am J Infect Control. 1987 Feb;15(1):1-6. doi: 10.1016/0196-6553(87)90069-1. PMID 3645972
- [Background] Iannini PB, Crossley K. Therapy of Staphylococcus aureus bacteremia associated with a removable focus of infection. Ann Intern Med. 1976 May;84(5):558-60. doi: 10.7326/0003-4819-84-5-558. PMID 1275357
- [Background] Jensen AG, Wachmann CH, Espersen F, Scheibel J, Skinhoj P, Frimodt-Moller N. Treatment and outcome of Staphylococcus aureus bacteremia: a prospective study of 278 cases. Arch Intern Med. 2002 Jan 14;162(1):25-32. doi: 10.1001/archinte.162.1.25. PMID 11784216
- See also: Related Info — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm